CLINICAL TRIAL: NCT01689727
Title: A Clinical Study to Evaluate the Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Subjects With Pituitary Tumors
Brief Title: Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Subjects With Pituitary Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.7
Record Dates: First submitted 2012-09-09; First posted 2012-09-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-09

CONDITIONS: Pituitary Tumors
Keywords: Pituitary Tumors
MeSH Terms: conditions — Pituitary Neoplasms

ARMS (1):
- Technetium Tc 99m EC20 (Other)
  Interventions: Drug: Technetium Tc 99m EC20

INTERVENTIONS:
Drug: Technetium Tc 99m EC20

SUMMARY:
Many types of cancers overexpress a receptor for the vitamin folate (Folate Receptor). This Phase 2 study will utilize a standard imaging radionuclide, technetium-99m, conjugated to a ligand (EC20) designed to bind to the folate receptor. The study is designed as an open-label, baseline-controlled study.

DETAILED DESCRIPTION:
This is a Phase 2 open-label, single-treatment group, baseline-controlled study designed to verify product safety, gather data on the percentage of subjects with pituitary tumors with increased uptake of FolateScan in tumors and correlate the immunohistochemical staining findings with the FolateScan images, in subjects with pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following eligibility requirements to be enrolled in the study:

1. Subject must be 18 years of age or older.
2. Subject must have a pituitary tumor.
3. Subject must have good kidney function.

3. Subject must provide written informed consent prior to enrollment.

Exclusion Criteria:

Subjects must be excluded if any of the following conditions are present:

1. Subject is pregnant or breastfeeding.
2. Subject is simultaneously participating in another investigational drug study.
3. Subject has completed the follow-up phase of any previous study loess than 30 days prior to enrollment in this study.
4. Subject is unable to tolerate conditions for radionuclide imaging.
5. Subject has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-09; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Oyesiku, MD, Principal Investigator — Emory Hospital
Locations (1):
- Emory Hospital, Atlanta, Georgia, United States